CLINICAL TRIAL: NCT04646369
Title: The Center for Enhancing Treatment & Utilization for Depression and Emergent Suicidality Phase 2-Study 1-Screening Wizard
Brief Title: Screening Wizard- Phase 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Kaiser Foundation Research Institute (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Oliver Lindhiem, Associate Professor of Psychiatry, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: STUDY20060325; P50MH115838-02 (NIH)
Record Dates: First submitted 2020-11-20; First posted 2020-11-27 (Actual); Results first posted 2022-09-27 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Depression; Suicidal Ideation
Keywords: depression; anxiety; suicidal ideation; treatment; referral; screening
MeSH Terms: conditions — Depression; Suicidal Ideation; Anxiety Disorders | interventions — Mass Screening

STUDY DESIGN:
Intervention Model Description: This study will use a parallel study design, where participants are randomized into three intervention groups ("screening as usual", Screening Wizard 2.0, Screening Wizard 2.0 + SOVA) and will receive interventions in parallel.
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors will be masked to the intervention condition at follow-up assessment time points.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- "screening as usual" (Active Comparator): Participants in the "screening as usual' group will have a symptoms scores report of results sent to their provider based on their Screening Wizard responses.
  Interventions: Behavioral: "screening as usual"
- Screening Wizard 2.0 (Experimental): Participants in the Screening Wizard 2.0 Report group will have a symptoms scores report of results and treatment preferences, barriers, and recommendations sent to their provider based on their Screening Wizard responses.
  Interventions: Behavioral: Screening Wizard 2.0
- Screening Wizard 2.0 + SOVA (Experimental): Participants in the Screening Wizard 2.0 + SOVA group will have a symptoms scores report of results and treatment preferences, barriers, and recommendations sent to their provider based on their Screening Wizard responses. This group will also receive access to the SOVA website aimed at addressing perceptions about mental health providing support to teens through peer interaction.
  Interventions: Behavioral: Screening Wizard 2.0 + SOVA

INTERVENTIONS:
Behavioral: "screening as usual" — Participants in this group will receive usual care at their pediatric primary care practice following information, psychoeducation, and referral to a mental health treatment provider
  Arms: "screening as usual"
Behavioral: Screening Wizard 2.0 — Screening Wizard is a decision support tool to guide the primary care provider to make a referral that reflects patient clinical needs and patient and parental treatment preferences and perceived barriers to treatment.
  Arms: Screening Wizard 2.0
Behavioral: Screening Wizard 2.0 + SOVA — Screening Wizard is a decision support tool to guide the primary care provider to make a referral that reflects patient clinical needs and patient and parental treatment preferences and perceived barriers to treatment. SOVA is a peer-support website that social workers and doctors moderate on a 24 hour a day basis.
  Arms: Screening Wizard 2.0 + SOVA

SUMMARY:
Screening Wizard (SW). Primary Care Providers (PCPs) are often uncertain about how to best refer adolescents who screen positive for depression or suicidality. Screen-positive youth who are either not in treatment, or express dissatisfaction with current treatment will be consented by an on-site research assistant (RA). Participants will answer questions via adaptive screens developed in a previous NIMH study (MH100155) for suicidal risk, anxiety, and mania. These will address perceived barriers and preferences about treatment. Participants are then randomized into 1 of 3 groups: 1) Providing the symptoms scores report of results to their provider based on their Screening Wizard responses (Screening as Usual); 2) Providing the symptoms scores report and their responses to treatment preferences and barriers including treatment recommendations their provider might suggest (Screening Wizard 2.0); or 3) Providing the report with treatment recommendations to their provider and a website called SOVA or Supporting Our Valued Adolescent, that is aimed at addressing perceptions about mental health providing support to teens through peer interaction that social workers and doctors moderate on a 24 hour a day basis (Screening Wizard 2.0 + SOVA).

DETAILED DESCRIPTION:
Screening Wizard will be delivered by Primary Care Providers (PCPs) at well child visits, beginning with screening occurring within the waiting room which will yield decision support guidance delivered and followed by the PCP at the same visit.

Assignment of Interventions: This study will randomize participants to one of three conditions in a 2:2:1 randomization scheme to either receive "screening as usual" (n=20), Screening Wizard 2.0 (n=40), or Screening Wizard 2.0 + SOVA (n =40)

Hypothesis: H1: Screening Wizard 2.0 will result in more referrals compared to "screening as usual" (increase >30% compared to "screening as usual")

H2: Screening Wizard 2.0 will result in higher rates of follow-through with mental health services compared to "screening as usual" (increase >30% compared to "screening as usual")

H3: Screening Wizard 2.0 will have higher adolescent and parent perception of being involved in a shared decision-making process compared to "Treatment as usual" (SW involvement > "screening as usual" involvement )

H4: Adolescent and parents in Screening Wizard 2.0 + SOVA will have less negative attitudes about psychotherapy, higher depression literacy, and a higher readiness for treatment as compared to Screening Wizard 2.0 alone or "screening as usual"

H5: Adolescent and parents in Screening Wizard 2.0 + SOVA will result in higher rates of follow-through with mental health services (defined as attendance at an initial appointment) compared to Screening wizard 2.0 alone (increase >10%) and "screening as usual" (increase >40%)

ELIGIBILITY:
Inclusion Criteria:

1. Youth aged 12-26yo
2. Biological or adoptive parent is willing to provide informed consent for teen to participate
3. Youth speaks and understands English

Exclusion Criteria:

1. Non English speaking
2. No parent willing to provide informed consent
3. Is currently experiencing acute mania or psychosis, evidence of an intellectual or developmental disorder (IDD), life threatening medical condition that requires immediate treatment, or other cognitive or medical condition preventing youth from understanding study and/or participating.

Ages: 12 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2021-09-17 (Actual); Study Completion 2021-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Lindhiem, PhD, Principal Investigator — University of Pittsburgh; Ana Radovic, Study Director — University of Pittsburgh
Locations (2):
- United States (2):
  - UPMC Center for Adolescent and Young Adult Health, Pittsburgh, Pennsylvania
  - Kids Plus Pediatrics, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
All requests for study data will follow NIMH's data sharing and data use policies. The final completely de-identified dataset(s) will include demographic and clinical data at baseline, and primary and secondary outcomes for all studies, including those funded by the innovation contests. These analytic datasets may also include derived variables with documentation. Our form datasets will include original case report forms, a detailed codebook of variable names, value labels, and programming formats and all study documentation including the protocol and manual of procedures. For descriptive/raw data, study investigators/study staff will upload to NIMH's National Database for Clinical Trials Related to Mental Health Illness (NDCT) on a semi-annual basis all analyzed data being uploaded prior to primary paper publication.
Time Frame: These data will be released to the NDCT soon after each project's "main outcomes" manuscript is accepted for publication
Access Criteria: In addition to public access to the NDCT, data can also be accessed by contacting ETUDES Center investigators.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | "Screening as Usual" | Screening Wizard 2.0 | Screening Wizard 2.0 + SOVA
Started | 23 | 38 | 39
Completed | 23 | 38 | 39
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | "Screening as Usual" | Screening Wizard 2.0 | Screening Wizard 2.0 + SOVA | Total
Number analyzed (Participants) | 23 | 38 | 39 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 15 | 10 | 29
  Between 18 and 65 years | 19 | 23 | 29 | 71
  >=65 years | 0 | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 1 | 3 | 3 | 7
  Female | 16 | 24 | 27 | 67
  Male to Female Transgender | 1 | 4 | 2 | 7
  Female to Male Transgender | 4 | 3 | 3 | 10
  Non Binary/Queer | 0 | 3 | 3 | 6
  Other | 1 | 1 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 2 | 5
  Not Hispanic or Latino | 19 | 38 | 37 | 94
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 7 | 10 | 23
  White | 16 | 26 | 21 | 63
  More than one race | 0 | 2 | 7 | 9
  Unknown or Not Reported | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Referred to Treatment
Description: The rate of personalized referrals by primary care providers and treatment initiation among adolescents who screen positive for depression or suicidal ideation will be monitored to determine if provider made referrals.
Time Frame: Baseline (in office) visit
Population: 92 of 100 participants had documentation or an accessible electronic medical record to review referrals made following screening wizard report. Note-Screening Wizard arm (N=38) and Screening Wizard + Sova arm (N=39) are combined because both arms received same Screening Wizard intervention but the 3rd Arm also received SOVA.
  Data was reviewed and entered from the electronic health record based on referrals made by pediatric providers at time the intervention was implemented.
Measure: Count of Participants; unit: Participants
Arm/Group | "Screening as Usual" | Screening Wizard 2.0
Number analyzed (Participants) | 22 | 70
Participants
  Drug or alcohol treatment services Referral | 0 | 1
  Emergency department services Referral | 0 | 0
  Family-based services Referral | 0 | 1
  In-home services Referral | 0 | 0
  Inpatient services Referral | 0 | 0
  Intensive Outpatient Program Referral | 0 | 1
  Outpatient psychotherapy/counseling Referral | 4 | 19
  Partial hospitalization Referral | 0 | 0
  Residential treatment facility Referral | 0 | 0
  School-based services Referral | 0 | 0
  Other Referral | 1 | 2

2. Secondary Outcome: Cost Analysis: Cost of Screening Wizard Intervention at Baseline
Description: An overall average of the cost of implementing the Screening Wizard intervention (including labor, equipment, supplies, facilitates) will be estimated at Baseline.
Time Frame: At Baseline visit
Population: Only participants who engaged in the Screening Wizard intervention are able to be analyzed for cost estimate. Both the "Screening Wizard 2.0 Report Group" arm and the Screening Wizard + SOVA Arm are included in this analysis. The intervention cost is only calculated for the intervention itself, not in the context of use of other services such as SOVA or those in the control group who may access other services.
Measure: Mean (Full Range); unit: dollars per participant
Arm/Group | Screening Wizard 2.0
Number analyzed (Participants) | 77
dollars per participant | 160.34 [81.54 to 198.88]

3. Secondary Outcome: Usability & Satisfaction
Description: Satisfaction to Screening Wizard will be assessed through questions developed by investigators to understand experience with the program. Questions investigators have adapted from literature reviews on satisfaction include:
  If a friend were in need of a mental health referral, would you recommend Screening Wizard to him/her? (SCALE: No, definitely not-Yes, definitely/1-4)
  How satisfied are you with the amount of help you received? (SCALE: Very dissatisfied-Very satisfied/1-4)
  Have the services you received helped you to deal more effectively with your problems? (SCALE: Seemed to make things worse-Yes, a great deal/1-4)
Time Frame: At exit interview after Baseline phone visit. The Baseline visit occurs 24-48 hours after initial screening and the exit interview call will be made within 1 month following the completion of the Baseline phone assessment
Population: All participants who reported to usability & satisfaction questions were analyzed from the 2 arms that used the Screening Wizard intervention. Note=Screening As Usual/Treatment As Usual (TAU) participants did not receive the items because they did not receive the intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Screening Wizard 2.0 | Screening Wizard 2.0 + SOVA
Number analyzed (Participants) | 38 | 39
score on a scale
  If a friend needed to talk to provider about emotional or mental health concerns would you recommend | 2.88 (0.7) | 2.89 (0.69)
  How satisfied with the amount of help you received? | 3.42 (0.5) | 3.39 (0.55)
  Have the services you received helped you to deal more effectively with your problems? | 2.94 (0.76) | 2.71 (0.75)

4. Secondary Outcome: Satisfaction With Technical Components
Description: Satisfaction with the technical components of interventions will be assessed through the certain questions from the Post System Satisfaction and Usability Questionnaire (PSSUQ). The PSSUQ is 19 items with response options ranging from 1 to 7 where 1= strongly disagree and 7= strongly agree. The PSSUQ has sub-scores derived from subsets of the questions which reflect system usefulness, information quality, and interface quality. 4 Questions from sub-domains were chosen to tailor the questioning to this particular intervention.
Time Frame: At exit interview after Baseline phone visit. The Baseline visit occurs 24-48 hours after initial screening and the exit interview call will be make within 1 month following the completion of the Baseline phone assessment
Population: All participants who reported to usability & satisfaction questions were analyzed from the 2 arms that used the Screening Wizard intervention. Note=TAU participants did not receive the items because they did not receive the intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Screening Wizard 2.0 | Screening Wizard 2.0 + SOVA
Number analyzed (Participants) | 38 | 39
score on a scale
  Overall, I am satisfied with how easy it is to use Screening Wizard | 6.41 (0.84) | 6.5 (0.83)
  Information such as online help, on-screen messages, other documentation...was clear | 6.13 (1.45) | 6.37 (1.13)
  I liked interacting with the Screening Wizard app | 5.81 (1.38) | 5.68 (1.3)
  needed to learn a lot of things before I could get going with the Screening Wizard | 1.22 (0.49) | 1.35 (0.95)

ADVERSE EVENTS:
Time Frame: participants were assessed for adverse events at each timepoint (baseline and 12 week follow-up)
Arm/Group | "Screening as Usual" | Screening Wizard 2.0 | Screening Wizard 2.0 + SOVA
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/38 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/38 | 0/39
Other Adverse Events (participants affected / at risk) | 0/23 | 0/38 | 0/39

LIMITATIONS AND CAVEATS:
The small sample limited the ability to detect statistical significance and practice sites had significant involvement from the research team. Both of these factors limit the generalizability of the results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-21): https://cdn.clinicaltrials.gov/large-docs/69/NCT04646369/Prot_SAP_001.pdf
  • Informed Consent Form (2020-10-05): https://cdn.clinicaltrials.gov/large-docs/69/NCT04646369/ICF_002.pdf